CLINICAL TRIAL: NCT05153070
Title: Clinical and Biological Responses to Repeated Administration of Low-dose Interleukin-2 in Patients With Type 1 Diabetes and a Residual Insulin Secretion
Brief Title: Ciclosporin Followed by Low-dose IL-2 in Patients With Recently Diagnosed Type 1 Diabetes
Acronym: DF-IL2-REP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Iltoo Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P120142
Record Dates: First submitted 2021-04-16; First posted 2021-12-10 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Type 1 Diabetes
Keywords: Interleukin 2; Ciclosporin; Auto-immune disease; Diabetes; Regulatory T cells; Immune tolerance; Immunotherapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Cyclosporine

STUDY DESIGN:
Intervention Model Description: Single group during ciclosporin treatment and parallel group during ILT-101 treatment
Who Masked: Participant, Investigator
Masking Description: all participant receive the treatment with Ciclosporin and double Blind for the treatment with IL-2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ciclosporin/ILT-101 (Experimental): Ciclosporin during 2 months (for all patients) followed by ILT-101 during 10 months
  Interventions: Drug: Cyclosporin; Drug: ILT101
- Ciclosporin/placebo (Placebo Comparator): Ciclosporin during 2 months (for all patients) followed by placebo during 10 months
  Interventions: Drug: Cyclosporin; Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporin — • Ciclosporin: 5mg/kg, twice a day, oral, between Day 1 and Day 60
Drug: ILT101 — • ILT-101: 1MIU/day in a volume of 1 ml; subcutaneous injection every day during 5 consecutive days and then every week between Day 63 and Day 354.
  Arms: Ciclosporin/ILT-101
Drug: Placebo — • Placebo with an identical formulation and regimen of injections i.e. Subcutaneous injection every day (5 consecutive days) then then every week between Day 63 and Day 354.
  Arms: Ciclosporin/placebo

SUMMARY:
Type 1 diabetes (T1D) is caused by the destruction of insulin-producing cells by effector T cells (Teffs), due to a deficiency of regulatory T cells (Tregs).

Ciclosporin effectively blocks the Teffs and controls diabetes, but cannot be considered as a long-term treatment. Low-dose interleukin-2 (ld IL-2) activates and expands Tregs in humans.

Hence, Ld IL-2 in patients in whom the autoimmune process was blocked early by a short treatment (2 months) of cyclosporine should restore immune homeostasis and maintain some insulin production over the long term.

DETAILED DESCRIPTION:
Primary Objective :

Tregs' response profile, after 4 administrations of 1MIU/day of IL-2 (Day 63-66) in patients with recently diagnosed type 1 diabetes who have been treated with ciclosporin for 2 months.

Primary assessment criterion:

Change in Tregs values at D67 compared to D63 (post-ciclosporin values)

Secondary objectives and secondary assessment criteria:

* Change in residual insulin secretion

  * AUC plasma C-peptide concentration after a mixed meal tolerance test at Month 6 (Day 179), Month 12 (Day 361) and after treatment discontinuation at Month 18 (Day 536) and Month 24 (Day 719) compared to baseline;
  * Insulin requirement, HbA1c dosage and IDAA1c score at Month 3 (Day 88), Month 6 (Day 179), Month 9 (Day 270), Month 12 (Day 361) and after treatment discontinuation at Month 18 (Day 536) and Month 24 (Day 719) compared to baseline
* Change in Tregs values at Month 3 (Day 88), Month 6 (Day 179), Month 9 (Day 270), Month 12 (Day 361) and after treatment discontinuation at Month 18 (Day 536) and Month 24 (Day 719) compared to baseline and post-ciclosporin values (Day 63)
* Ciclosporin and ILT-101/placebo compliance
* Tolerance

Experimental design:

This is a monocentric, randomized, placebo controlled, double-blind trial in parallel-groups, evaluating a treatment by cyclosporine 7mg/kg/day during 2 months followed by ILT-101/placebo, 1 MIU daily for 5 days and 1 MIU every week, during 10 months.

Population involved:

Male or female, aged between 16 and 35 years, with recent diagnosis of type 1 diabetes (< 3 months).

Number of subjects: 24 Inclusion period: 12 months Duration of patient participation: 24 months (treatment period: 12 months, follow-up period: 12months) Total duration of the study: 37 months

ELIGIBILITY:
Inclusion Criteria:

* • Age at inclusion between ≥ 16 years old (Tanner 5 pubertal stage) and ≤ 45 years old

  * Type 1 diabetes according to ADA criteria, with at least 1 positive autoantibody among the following: anti-islet, anti-GAD, anti-IA2, anti-ZnT8 and anti-insulin.
  * Diagnosis ≤ 3 months
  * No acid ketosis
  * No weight loss > 10% OR with fasting C-peptide ≥ 0.1 nmol/L (after a period of ≥ 15 days following the initiation of insulin therapy
  * Absence of clinically significant biological abnormalities on hematological, biochemical, hepatic, renal and thyroid tests.
  * No documented history of heart disease, no family history of sudden death, AND normal ECG.
  * Effective contraception in men and women of childbearing potential > 2 weeks prior to first administration of the investigational drug and throughout the treatment period (if sexually active). Specifically for women of childbearing age and sexually active, they must use an effective contraceptive method (Pearl Index < 1). The following methods are acceptable: oral hormonal contraceptives, injectable, or implanted (with the exception of oral minipills: i.e. low doses of gestagens which are not acceptable (lynestrenol and norestisteron), intrauterine contraceptives (e.g. progestin-release systems)),
  * Free, informed and written consent, signed by the patient and the investigator, prior to any examination required by the trial.

If the patient is a minor, the signatures of both parents and of the child will be collected (or the legal representative if only one parent is alive).

Exclusion Criteria:

* Known contraindications to IL2 treatment:

  * Hypersensitivity to the active substance or to one of the excipients.
  * Signs of active infection requiring antibiotics
  * Documented history of clinical autoimmune disease
  * Oxygen saturation ≤ 90%
  * Existence of a serious dysfunction in a vital organ
  * History of organ allograft,
* Known contraindications to treatment with cyclosporine
* Presence of unauthorized treatment, i.e. cytotoxic drugs, products known for their impact on blood glucose levels or for their interactions with the treatments under trial
* Patients who have received anti-diabetic treatment other than insulin for more than 3 consecutive months.
* Anti-thyroperoxidase positive and abnormal TSH and T4 at inclusion
* Anti-transglutaminase positive at inclusion
* EBV viral load > 2000 IU/ml
* CMV viral load > 400 IU/ml
* HBV, HCV or HIV infection
* Lymphopenia ≤ 1000/ mm3
* Presence or history of cancer that has been cured for less than five years, except in situ cervical or basal cell carcinoma in early stage management,
* Participation in other intervention research involving humans < 3 months,
* Pregnant or breastfeeding women
* Lack of social security affiliation (as a beneficiary or assignee)
* Vaccination with live attenuated virus during the last 4 weeks before the start of the experimental treatment and during the entire treatment phase.
* Patient with active SARS-CoV-2 infection
* Patient with chronic respiratory disease
* Subject under legal protection (such as tutorship, curatorship, or judicial safeguard)
* Subject hospitalized without consent, unable to express consent or deprived of liberty

Ages: 16 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-04-21 (Estimated); Study Completion 2028-04-21 (Estimated)

PRIMARY OUTCOMES:
Treg variation | From Day 63 to Day 67
  Change in Tregs values at Day 67 compared to Day 63 (post-ciclosporin value)

SECONDARY OUTCOMES:
Change in Area under curve (AUC (T0-T120) of serum C-peptide at month 6 | up to month 6
  Change in Area under curve (AUC (T0-T120) of serum C-peptide after mixed-meal tolerance test compared to baseline
  2. Variation in HbA1c value (in %) 3. Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)].
  4. Change in Insulin requirement (insulin dose in international units per kilogram per 24 h 5. Change in Tregs values (in %/CD4+) at month 3, month 6, month 9, month 12 and after treatment interruption at month 18 and month 24 compared to baseline and post-cyclosporin values (Day 63)
Change in Area under curve (AUC (T0-T120) of serum C-peptide at month 12 | up to month 12
  Change in Area under curve (AUC (T0-T120) of serum C-peptide after mixed-meal tolerance test compared to baseline
  2. Variation in HbA1c value (in %) 3. Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)].
  4. Change in Insulin requirement (insulin dose in international units per kilogram per 24 h 5. Change in Tregs values (in %/CD4+) at month 3, month 6, month 9, month 12 and after treatment interruption at month 18 and month 24 compared to baseline and post-cyclosporin values (Day 63)
Change in Area under curve (AUC (T0-T120) of serum C-peptide at month 24 | up to month 24
  Change in Area under curve (AUC (T0-T120) of serum C-peptide after mixed-meal tolerance test compared to baseline
  2. Variation in HbA1c value (in %) 3. Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)].
  4. Change in Insulin requirement (insulin dose in international units per kilogram per 24 h 5. Change in Tregs values (in %/CD4+) at month 3, month 6, month 9, month 12 and after treatment interruption at month 18 and month 24 compared to baseline and post-cyclosporin values (Day 63)
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at day 63, | up to day 63
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 3 | up to month 3
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 6 | up to month 6
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 9 | up to month 9
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 12 | up to month 12
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 18 | up to month 18
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to Baseline at month 24 | up to month 24
  Variation in HbA1c value (in %) during the treatment period and during the 1-year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at day 63 | up to day 63
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period up to month 3 | up to month 3
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at month 6 | up to month 6
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at month 9 | up to month 9
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at month 12 | up to month 12
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at day month 18 | up to month 18
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Variation in IDAA1c scoreduring the treatment period and during the 1 year follow-up period at month 24 | up to month 24
  Variation in IDAA1c score (IDAA1c score = HbA1c (in %) + [4 × insulin dose (in international units per kilogram per 24 h)] during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at day 30 | up to day 30
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at day 63 | up to day 63
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 3 | up to month 3
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 6 | up to month 6
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 9 | up to month 9
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 12 | up to month 12
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 18 | up to month 18
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period at month 24 | up to month 24
  Change in Insulin requirement (insulin dose in international units per kilogram per 24 h) during the treatment period and during the 1 year follow-up period compared to baseline
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at day 30 | up to day 30
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at day 63 | up to day 63
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 3 | up to month 3
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 6 | up to month 6
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 9 | up to month 9
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 12 | up to month 12
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 18 | up to month 18
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
Change in Tregs values (in %/CD4+) after treatment interruption and post-cyclosporin values at month 24 | up to month 24
  Change in Tregs values (in %/CD4+) after treatment interruption compared to baseline and post-cyclosporin values
incidence of adverse events at day 30 | up to day 30
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at day 63 | up to day 63
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 3 | up to month 3
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 6 | up to month 6
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 9 | up to month 9
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 12 | up to month 12
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 18 | up to month 18
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24
incidence of adverse events at month 24 | up to month 24
  incidence of adverse events throughout the study (according to NCI-CTC AE classification) to the Baseline to month 24

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, MD, Ph.D, Study Director — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS; Agnès Hartmann, MD, Ph.D, Principal Investigator — APHP(ASSISTANCE PUBLIQUE DES HOPITAUX DE PARIS
Locations (1):
- Lorenzon Roberta, Paris, France

IPD SHARING:
Plan to Share IPD: No